CLINICAL TRIAL: NCT01815554
Title: Long-term Follow-up of Patients With Ventilatory Dependent High Tetraplegia Managed With Diaphragmatic Pacing Systems
Brief Title: Follow up Study of Diaphragm Pacing for Patients With High Tetraplegia
Status: Completed | Type: Observational
Sponsor: Craig Hospital (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 133N110006
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Tetraplegia; Spinal Cord Injury
Keywords: Tetraplegia; Spinal Cord Injury; Ventilator; Diaphragmatic Pacing System
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DPS Cohort: All patients implanted with a DPS within the past 5 years at one of 6 collaborating sites will be included. Patients will be interviewed as they cross their 1st, 3rd, 5th or 7th anniversary with the DPS.

SUMMARY:
This is an observational longitudinal study designed to identify and describe long term outcomes for patients with high tetraplegia who use a Diaphragmatic Pacing System (DPS). As this is not a randomized or experimental study, no specific hypotheses are proposed. The data collected will enable us to answer the following research questions:

1. What are the patterns of long-term DPS use (hours per day using DPS, changes in DPS stimulus parameters, abandonment of DPS and related reasons).
2. What mechanical problems have DPS users encountered (system failure, repairs needed)?
3. What are the frequency of and reasons for rehospitalization following DPS implant?
4. What levels of care are needed at home to manage the DPS?
5. How do DPS users feel about the system (satisfaction, comfort, vocalization, taste, swallowing)?

DETAILED DESCRIPTION:
Ventilatory dependent high tetraplegia is a relatively rare but devastating condition. Review of National Spinal Cord Injury Database statistics show that only 3.6% of patients with tetraplegia are ventilator dependent at one year post injury.1 A subset of individuals who are ventilatory dependent in the long term and have upper motor neuron paralysis of the diaphragm are candidates for electrophrenic respiration (EPR) which can create inspiratory function through electrical stimulation of the phrenic nerves, resulting in diaphragmatic contraction. The use of this technology in ventilatory dependent tetraplegia was first described almost 40 years ago with a pacing system using cuff electrodes surgically placed around the phrenic nerve in the neck.2 The concept of EPR via minimally invasive laparoscopically placed diaphragmatic electrodes was first reported in 2002.3 This new Diaphragmatic Pacing System (DPS) had the distinct advantage of requiring less invasive surgery for electrode implantation compared to the phrenic cuff electrode system which required surgical exploration of the neck. In some settings, the DPS system has been implanted as an outpatient surgery. The DPS had a potential disadvantage however in that, unlike the traditional EPR system, the stimulating electrode leads are externalized posing an infection risk and the electrodes are attached to a moving muscle creating a risk for dislodgement. Once the system achieved FDA Humanitarian Use Device (HUD) exemption status in 2008, there was adoption of the Diaphragm Pacing System (DPS) among a number of SCI centers as a treatment option for patients with ventilatory dependent high tetraplegia. Reporting of long-term outcomes of DPS in the SCI population is limited to a 2009 report authored by the system inventor on 50 patients with average follow-up of 2.0 ± 1.5 years (median 1.6 years, range 0.5-8.0 years).4 The six SCIMS centers participating in this module research propose to collect long-term follow-up data on DPS patients implanted and/or followed at their centers since 2007. This project will enable the reporting of independent long-term utilization, effectiveness, satisfaction, durability and safety outcomes of this innovative technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously incurring a traumatic spinal cord injury resulting in high tetraplegia
* Patients implanted with DPS

Exclusion Criteria:

* Implementation of DPS prior to 2003

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals implanted with DPS since 2003 who are being followed at one of the 6 collaborating study sites, including individuals who undergo DPS implantation during the funding cycle through October of 2014. Currently, there are approximately 60 individuals who comprise the existing clinical cohort of eligible participants. Individuals who are implanted during the funding cycle also will be eligible for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Long-term utilization, effectiveness, satisfaction, durability and safety of implanted Diaphragmatic Pacing Systems | 1 year anniversary of original implemenation date
  Patients implanted with a DPS within the past 5 years will be included in this study. Telephone or in-person interviews will be conducted with the above individuals as they cross their 1st, 3rd, 5th, or 7th anniversary with the DPS system. All individuals are expected to complete at least 2 interviews during the study period.
Long-term utilization, effectiveness, satisfaction, durability and safety of implanted Diaphragmatic Pacing Systems | 3 year anniversary of original implemenation date
  Patients implanted with a DPS within the past 5 years will be included in this study. Telephone or in-person interviews will be conducted with the above individuals as they cross their 1st, 3rd, 5th, or 7th anniversary with the DPS system. All individuals are expected to complete at least 2 interviews during the study period.
Long-term utilization, effectiveness, satisfaction, durability and safety of implanted Diaphragmatic Pacing Systems | 5 year anniversary of original implemenation date
  Patients implanted with a DPS within the past 5 years will be included in this study. Telephone or in-person interviews will be conducted with the above individuals as they cross their 1st, 3rd, 5th, or 7th anniversary with the DPS system. All individuals are expected to complete at least 2 interviews during the study period.
Long-term utilization, effectiveness, satisfaction, durability and safety of implanted Diaphragmatic Pacing Systems | 7 year anniversary of original implemenation date
  Patients implanted with a DPS within the past 5 years will be included in this study. Telephone or in-person interviews will be conducted with the above individuals as they cross their 1st, 3rd, 5th, or 7th anniversary with the DPS system. All individuals are expected to complete at least 2 interviews during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States